CLINICAL TRIAL: NCT05868954
Title: Implementation of a Mediterranean Diet Program for Overweight or Obese Pregnant Women in a Low-resource Clinical Setting
Acronym: MedDiet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00096969; UL1TR001420 (NIH)
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-03

CONDITIONS: Gestational Weight Gain; Diet, Healthy
Keywords: Mediterranean Diet; Overweight; Pregnant Women; Obese
MeSH Terms: conditions — Gestational Weight Gain; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- American College of Obstetricians and Gynecologists (ACOG)-based Dietary Program (Active Comparator): Routine dietary counseling program
  Interventions: Behavioral: ACOG-based Dietary Program
- Mediterranean Diet (MedDiet) Program (Experimental): Well-known healthy diet that consists of a large amount of plant-based foods such as fruits, vegetables, beans, and nuts with extra virgin olive oil (EVOO) as the principal source of fat. Dairy, fish, and poultry are consumed in moderation and red meat only eaten occasionally.
  Interventions: Behavioral: MedDiet Program

INTERVENTIONS:
Behavioral: MedDiet Program — Subjects allocated to the MedDiet Program group will receive counseling based on the principles of the traditional MedDiet with a focus on a general change in diet instead of micronutrients or macronutrients. Diet adherence will be assessed using a 14 question questionnaire. Participants will receive 6, free traditional MedDiet meals every 3 weeks between enrollment and until the subject is approximately 38 weeks pregnant. In addition, participants will receive olive oil and nuts during their enrollment visit and during their routine 26-30 week prenatal visit.
  Arms: Mediterranean Diet (MedDiet) Program
Behavioral: ACOG-based Dietary Program — Following ACOG recommendation, subjects allocated to the ACOG-based Dietary Program group, will receive routine counseling on healthy eating. This will include advice on the consumption of grains, fruits, vegetables, protein, and dairy foods recommended during pregnancy. Diet adherence will be assessed using an 18 question questionnaire. Participants will receive 6, free traditional healthy meals every 3 weeks between enrollment and until the subject is approximately 38 weeks pregnant. In addition, participants will receive canola oil and healthy snacks during their enrollment visit and during their routine 26-30 week prenatal visit.
  Arms: American College of Obstetricians and Gynecologists (ACOG)-based Dietary Program

SUMMARY:
The purpose of this Pilot randomized clinical Trial is to compare two healthy diet styles during pregnancy. Patients between 8 and 16 weeks of gestation who agree to participate will be randomly assigned (like flipping a coin) to either receive routine healthy diet advice and counseling, or to receive advice and counseling for the Mediterranean style diet. Our current routine healthy diet program follows the recommendations provided by the American College of Obstetricians and Gynecologists (ACOG). It recommends the consumption of grains, fruits, vegetables, protein foods, and dairy foods during pregnancy. The Mediterranean diet (MedDiet) is a well-known healthy diet that consists of a large amount of plant-based foods such as fruits, vegetables, beans, and nuts with olive oil as the principal source of fat. Dairy, fish, and poultry are consumed in moderation and red meat only eaten occasionally. Throughout their pregnancy, participants will receive free food and be assessed to determine adherence to the diet and receive counseling to reinforce diet recommendations.

DETAILED DESCRIPTION:
The Mediterranean diet (MedDiet) is a well-known healthy diet that consists of a large amount of plant-based foods such as fruits, vegetables, beans, and nuts with extra virgin olive oil (EVOO) as the principal source of fat. Dairy, fish, and poultry are consumed in moderation and red meat only eaten occasionally. A growing body of evidence demonstrates that outside of pregnancy, the MedDiet is associated with a reduction of cardiovascular disease, diabetes, metabolic syndrome, and certain cancers. However, the potential clinical benefits of MedDiet in pregnancy are understudied with most data originating from clinical trials in Europe. Proper nutrition during pregnancy has multiple health benefits. A mother eating a healthy diet has a higher probability of meeting the demands required for a normal fetal development. In addition, she is more likely to achieve the recommended gestational weight gain thereby reducing the risk of pregnancy-related complications. Finally, a healthy diet is associated with a reduction of chronic conditions such as cardiovascular disease and diabetes later in life for both the mother and the infant.

ELIGIBILITY:
Inclusion Criteria:

* Viable singleton pregnancy in the first trimester (6 0/7- 16 6/7 weeks); includes twins reduced to singleton spontaneously or vanishing twin syndrome
* BMI ≥ 25.0 kg/m2; calculated by dividing maternal weight in kilograms by height in meters squared using a calibrated scale and standard metric measure
* Confirmed intrauterine pregnancy by ultrasound exam (6-16 weeks)
* Age 18 years or older
* Primary language of English or Spanish

Exclusion Criteria:

* BMI < 25.0 kg/m2
* Known pre-pregnancy diabetes
* Hemoglobin glycosylated (A1C) > 5.7% at first prenatal visit
* Pre-pregnancy hypertensive disease
* Non-viable pregnancy
* Known allergies to an essential component(s) of MedDiet
* Inability to read or write in primary language
* Mental incapacity to make medical decisions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Viable singleton pregnancy
Enrollment: 41 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Mateus Nino, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Myers Park OB/GYN, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program: Routine dietary counseling program
  ACOG-based Dietary Program: Following ACOG recommendation, subjects allocated to the ACOG-based Dietary Program group, will receive routine counseling on healthy eating. This will include advice on the consumption of grains, fruits, vegetables, protein, and dairy foods recommended during pregnancy. Diet adherence will be assessed using a 14 question questionnaire. Participants will receive 6, free traditional healthy meals every 3 weeks between enrollment and until the subject is approximately 38 weeks pregnant. In addition, participants will receive canola oil and healthy snacks during their enrollment visit and during their routine 26-30 week prenatal visit.
- Mediterranean Diet (MedDiet) Program: Well-known healthy diet that consists of a large amount of plant-based foods such as fruits, vegetables, beans, and nuts with extra virgin olive oil (EVOO) as the principal source of fat. Dairy, fish, and poultry are consumed in moderation and red meat only eaten occasionally.
  MedDiet Program: Subjects allocated to the MedDiet Program group will receive counseling based on the principles of the traditional MedDiet with a focus on a general change in diet instead of micronutrients or macronutrients. Diet adherence will be assessed using an 18 question questionnaire. Participants will receive 6, free traditional MedDiet meals every 3 weeks between enrollment and until the subject is approximately 38 weeks pregnant. In addition, participants will receive olive oil and nuts during their enrollment visit and during their routine 26-30 week prenatal visit.
Period: Overall Study
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Started | 21 | 20
Completed | 18 | 15
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Participant delivered | 1 | 1
Not completed — Miscarriage | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.24 (5.36) | 26.86 (5.32) | 28.59 (5.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 20 | 39
  Not Hispanic or Latino | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Diet Adherence Assessment Scores Continuous
Description: The Routine Healthy Diet Assessment Questionnaire consists of 15 items. Each item is scored as 1 for adherence and 0 for non-adherence, with some items having trimester-specific scoring. The total score is the sum of all items, ranging from 0 (no adherence) to 15 (full adherence). Higher scores indicate better adherence to the routine healthy diet .The MedDiet Assessment Questionnaire consists of 17 items. Each item is scored as 1 for adherence and 0 for non-adherence. The total score is the sum of all items, ranging from 0 (no adherence) to 17 (full adherence). Higher scores indicate better adherence to the Mediterranean diet.
Time Frame: week 38
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
score on a scale | 9.0 [7.5 to 10.0] | 11 [10.0 to 13.0]

2. Secondary Outcome: Gestational Weight Gain (GWG)
Description: Total GWG will be calculated by subtracting the participant's weight (lbs.) at the initial prenatal visit from the weight (lbs.) at time of the delivery or at the last prenatal visit. GWG in the first trimester (6-13 weeks), second trimester (14-26 weeks), and third trimester (27-40 weeks) will also be calculated. Calibrated weight scales will be used at our clinic and at the hospital. Compliance rate of GWG based on Institute of Medicine (IOM) guidelines for overweight and obese women will be compared between the MedDiet and the control group.
Time Frame: week 40
Measure: Mean (Standard Deviation); unit: pounds
Groups:
- American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program: Routine dietary counseling program
  ACOG-based Dietary Program: Following ACOG recommendation, subjects allocated to the ACOG-based Dietary Program group, will receive routine counseling on healthy eating. This will include advice on the consumption of grains, fruits, vegetables, protein, and dairy foods recommended during pregnancy. Diet adherence will be assessed using a questionnaire. Participants will receive 6, free traditional healthy meals every 3 weeks between enrollment and until the subject is approximately 38 weeks pregnant. In addition, participants will receive canola oil and healthy snacks during their enrollment visit and during their routine 26-30 week prenatal visit.
- Mediterranean Diet (MedDiet) Program: Well-known healthy diet that consists of a large amount of plant-based foods such as fruits, vegetables, beans, and nuts with extra virgin olive oil (EVOO) as the principal source of fat. Dairy, fish, and poultry are consumed in moderation and red meat only eaten occasionally.
  MedDiet Program: Subjects allocated to the MedDiet Program group will receive counseling based on the principles of the traditional MedDiet with a focus on a general change in diet instead of micronutrients or macronutrients. Diet adherence will be assessed using a questionnaire. Participants will receive 6, free traditional MedDiet meals every 3 weeks between enrollment and until the subject is approximately 38 weeks pregnant. In addition, participants will receive olive oil and nuts during their enrollment visit and during their routine 26-30 week prenatal visit.
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
pounds | 24.07 (10.47) | 19.54 (8.51)

3. Secondary Outcome: Cardiometabolic Biomarkers - Hemoglobin A1C Levels
Description: Hypothesize that consuming the Mediterranean diet (MedDiet) may be associated with improved cardiometabolic biomarkers during pregnancy. Specifically, MedDiet might help reduce the physiological rise in lipids, enhance insulin sensitivity, and lower markers of subclinical inflammation, such as C-reactive protein (CRP). Pregnancy is usually marked by increased levels of total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), and triglycerides, especially in the second and third trimesters, along with increased insulin resistance. This study aims to determine whether MedDiet influences these biomarkers. Maternal lipid profiles, random glucose levels, hemoglobin A1C, and CRP will be measured at baseline (first or second trimester) and between 26-30 weeks of gestation among participants in both the intervention and control groups. Lab samples will be collected during routine blood draws for prenatal care.
Time Frame: Week 30
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
percentage | 5.10 [5.00 to 5.30] | 4.90 [4.80 to 5.25]

4. Secondary Outcome: Cardiometabolic Biomarkers - C-reactive Protein (CRP) Levels
Description: Consumption of MedDiet is associated with lower levels of total cholesterol, reduces insulin resistance preventing type 2 diabetes and Gestational diabetes mellitus (GDM), and reduces markers of subclinical inflammation such as C-reactive protein (CRP). Pregnancy is characterized by increased levels of total cholesterol, low-density lipoprotein (LDP), high-density lipoprotein (HDL), and triglycerides, especially in the second and third trimester, and pregnancy is a state of increased insulin resistance. There is limited knowledge about the effect of MedDiet on cardiometabolic biomarkers during pregnancy. Maternal lipid profile, random glucose level, hemoglobin A1C, and CRP levels will be compared at baseline (first or early second trimester) and at 26-30 weeks of gestation among participants in the intervention and the control groups. The labs will be obtained at the same time of scheduled blood draws for routine prenatal labs.
Time Frame: Week 30
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
mg/dL | 1.00 [0.40 to 1.50] | 0.90 [0.45 to 1.90]

5. Secondary Outcome: Cardiometabolic Biomarkers - Triglycerides
Description: as for outcome 4
Time Frame: Week 30
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
mg/dL | 217.66 (14.21) | 261.23 (36.27)

6. Secondary Outcome: Cardiometabolic Biomarkers - Glucose Level
Description: as for outcome 4
Time Frame: Week 30
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
mg/dL | 86 [82 to 97] | 98 [81 to 106]

7. Secondary Outcome: Cardiovascular Parameters - Blood Pressure (BP) Values (Diastolic)
Description: MedDiet is associated with reduction of blood pressure (BP) in non-pregnant adult overweight or obese women. Physiological changes of blood pressure (BP) during pregnancy are characterized by reduction of BP in the second trimester with return to the pre-pregnancy level late in the third trimester and postpartum period. Heart rate (HR) increases by 20% to 25% over baseline during gestation. Maternal BP and HR will be obtained by a calibrated automated oscillometric device during prenatal visits from the first to the third trimesters following the standardized technique established in our clinic. Trends of BP and HR throughout gestation will be compared among women allocated in the intervention and the control groups.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
mmHg | 69.87 (8.34) | 70.80 (9.90)

8. Secondary Outcome: Cardiovascular Parameters - Blood Pressure (BP) Values (Diastolic)
Description: as for outcome 7
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
mmHg | 67.20 (6.49) | 67.80 (11.91)

9. Secondary Outcome: Cardiovascular Parameters - Blood Pressure (BP) Values (Diastolic)
Description: as for outcome 7
Time Frame: Week 30
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
mmHg | 67.20 (6.09) | 66.60 (8.53)

10. Secondary Outcome: Cardiovascular Parameters - Blood Pressure (BP) Values (Diastolic)
Description: as for outcome 7
Time Frame: Week 38
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
mmHg | 73.93 (5.43) | 67.80 (10.06)

11. Secondary Outcome: Cardiovascular Parameters - Blood Pressure (BP) Values (Systolic)
Description: as for outcome 7
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
mmHg | 116.33 (9.34) | 116.27 (9.91)

12. Secondary Outcome: Cardiovascular Parameters - Blood Pressure (BP) Values (Systolic)
Description: as for outcome 7
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
mmHg | 113.13 (10.14) | 109.73 (12.40)

13. Secondary Outcome: Cardiovascular Parameters - Blood Pressure (BP) Values (Systolic)
Description: as for outcome 7
Time Frame: Week 30
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
mmHg | 114.00 (17.39) | 109.53 (12.21)

14. Secondary Outcome: Cardiovascular Parameters - Blood Pressure (BP) Values (Systolic)
Description: as for outcome 7
Time Frame: Week 38
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
mmHg | 118.13 (7.91) | 109.80 (10.44)

15. Other Pre Specified Outcome: Initial Heartrate
Description: as for outcome 7
Time Frame: Week 16
Population: Data not collected
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: Number of Adverse Pregnancy Outcomes - Gestational Hypertension, Pre-eclampsia, Eclampsia
Description: examine the most common Adverse Pregnancy Outcomes (APO) associated with overweight and obesity: preeclampsia, eclampsia, gestational hypertension, gestational diabetes mellitus, preterm birth, cesarean delivery, large for gestational age infant.
Time Frame: week 40
Measure: Number; unit: Number of events
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
Number of events | 5 | 2

17. Other Pre Specified Outcome: Number of Adverse Pregnancy Outcomes (APO) Gestational Diabetes Mellitus
Description: as for outcome 16
Time Frame: week 40
Measure: Number; unit: Number of events
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
Number of events | 3 | 5

18. Other Pre Specified Outcome: Number of Adverse Pregnancy Outcomes (APO) Preterm Birth
Description: as for outcome 16
Time Frame: week 36
Measure: Number; unit: Number of events
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
Number of events | 2 | 2

19. Other Pre Specified Outcome: Number of Adverse Pregnancy Outcomes (APO) Cesarean Delivery
Description: as for outcome 16
Time Frame: week 40
Measure: Number; unit: Number of events
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
Number of events | 7 | 6

20. Other Pre Specified Outcome: Number of Adverse Pregnancy Outcomes (APO) Large for Gestational Age Infant
Description: as for outcome 16
Time Frame: week 40
Measure: Number; unit: Number of events
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
Number analyzed (Participants) | 21 | 20
Number of events | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program | Mediterranean Diet (MedDiet) Program
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 8/21 | 7/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | American College of Obstetricians and Gynecologists (ACOG)-Based Dietary Program (N=21) | Mediterranean Diet (MedDiet) Program (N=20)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1)
Gestational diabetes mellitus (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/54/NCT05868954/Prot_SAP_001.pdf
  • Informed Consent Form (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT05868954/ICF_000.pdf